CLINICAL TRIAL: NCT03691558
Title: Effects of Five Weeks of Ketogenic Diet on Long Distance Triathletes Performance
Brief Title: Effects of Ketogenic Diet on Triathlon's Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Universidade Federal de Goias (Other); University of Palermo (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Associate Professor, University of Padova
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KDTRI17
Record Dates: First submitted 2018-05-15; First posted 2018-10-01 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Ketogenic Dieting; Physical Activity
Keywords: ketogenic diet; triathlon; VO2max; PPO
MeSH Terms: conditions — Motor Activity | interventions — Diet, Ketogenic; Diet, Western

STUDY DESIGN:
Intervention Model Description: It is single blind, parallel arms study
Who Masked: Outcomes Assessor
Masking Description: Treatment and control were masked with A and B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Experimental): Subjects followed 5 weeks of ketogenic diet
  Interventions: Other: Ketogenic diet
- Western Diet (Active Comparator): Subjects followed 5 weeks of a western diet
  Interventions: Other: Western Diet

INTERVENTIONS:
Other: Ketogenic diet — total daily caloric intake was divided into 5 meals. Individual daily caloric need is calculated referring to body composition and adjusted for daily activity (Frankenfield, Roth-Yousey, & Compher, 2005; Wang et al., 2000). Macronutrients percentage is 68% fat, 26% protein and 6% carbohydrate Paoli et al. 2013). Very low carbohydrate foods that simulate carbohydrates taste food like croissants, bread and cracked slices made by Le Gamberi Foods (Forlì, Italy), are used for a better compliance to the dietary intervention
  Arms: Ketogenic diet
Other: Western Diet — total daily caloric intake was divided into 5 meals. Individual daily caloric need is calculated referring to body composition and adjusted for daily activity (Frankenfield, Roth-Yousey, & Compher, 2005; Wang et al., 2000). The diet macronutrient percentage distribution is the following: protein is 25% of TDC (total daily calories), fat is 20% of TDC and carbohydrates represented the 55% of TDC
  Arms: Western Diet

SUMMARY:
The study aimed to verify the effects of 5 weeks of ketogenic diet (KD) on some performance index in long distance triathletes

DETAILED DESCRIPTION:
16 well trained male long distance Triathletes participates in the study (30.65 ± 10.77 years of age), with minimum one year of triathlon competition experience and 8-10 hours of training per week. All subjects had a personal interview made by a registered Medical Doctor about the diet intervention prior to the beginning of the study. Moreover participants were educated about the benefits and limitations of the two different dietary treatments and asked to nominate their preference for, or non-acceptance of, each of these interventions. Thus participants also decided liberally if participate for the diet intervention or not. This choice was decided to prevent any type of dropout in the KD group, considering that a free and conscious choices is better for the adherence on a strict diet like ketogenic diet . Investigators were thus able to allocate the athletes to their preferred treatment, while achieving suitable matching of groups based on age, body mass and aerobic power. All the participants were healthy and injured free, and not consuming a low carbs diet prior to the study. The diet macronutrient percentage distribution was the following: for ND the percentages were 25% of TDC (total daily calories), fat were 20% of TDC and carbohydrates represented the 55% of TDC; for KD the percentages were 68% fat, 26% protein and 6% carbohydrate. In the KD very low carbohydrate foods that simulate carbohydrates taste food like croissants, bread and cracked slices made by Le Gamberi Foods (Forlì, Italy), were used for a better compliance to the dietary intervention. Subjects undertaken an anthropometric test and two different cardiopulmonary tests with a professional cycloergometer (MARCA). The anthropometric measures were taken to evaluated body weight. height and body composition . After the body composition analysis subjects underwent to a maximal cardiopulmonary test (GXT) to evaluate the maximal oxygen consumption (VO2max). The following day subjects performed 60 minutes at 45% of PPO to assess endurance performance at ironman biking race-pace. The day after test session KD group started the KD 5 weeks. The Control Group (S) followed his habitual normo-caloric, balanced diet. The same order and procedures were conducted for testing the subjects post diet intervention. Anthropometric and performance test was conducted in the same order for each subjects and at the same time of the day. Blood ketones were measured each other day to ensure the compliance to KD

ELIGIBILITY:
Inclusion Criteria:

* long distance Triathletes (8-10 hours of training per week), competing in half Ironman or Ironman
* no previous experience of low carbohydrate diet
* more than 3 years of training

Exclusion Criteria:

* recent (less than 6 months) musculoskeletal injuries
* more than 2 months without training in the last 2 years

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
VO2 at 45% of peak power output | after 5 weeks
  We measured the mean VO2 during one hour at the 45% of peak power output (PPO) measured during the first test

SECONDARY OUTCOMES:
VO2 per Kg/bw | after 5 weeks
  VO2 measured as ml O2 per kilograms of body weight
VO2max | after 5 weeks
  Maximal oxygen consumption measured through a incremental bike test
Body composition LBM | after 5 weeks
  Lean body mass (Kg) measured by Body Impedence Analysis
Body composition FM | after 5 weeks
  Fat mass (Kg) measured by Body Impedence Analysis
Body Weight | after 5 weeks
  in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — DSB University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wroble KA, Trott MN, Schweitzer GG, Rahman RS, Kelly PV, Weiss EP. Low-carbohydrate, ketogenic diet impairs anaerobic exercise performance in exercise-trained women and men: a randomized-sequence crossover trial. J Sports Med Phys Fitness. 2019 Apr;59(4):600-607. doi: 10.23736/S0022-4707.18.08318-4. Epub 2018 Apr 4. PMID 29619799
- [Background] Carr AJ, Sharma AP, Ross ML, Welvaert M, Slater GJ, Burke LM. Chronic Ketogenic Low Carbohydrate High Fat Diet Has Minimal Effects on Acid-Base Status in Elite Athletes. Nutrients. 2018 Feb 18;10(2):236. doi: 10.3390/nu10020236. PMID 29463034
- [Background] McSwiney FT, Wardrop B, Hyde PN, Lafountain RA, Volek JS, Doyle L. Keto-adaptation enhances exercise performance and body composition responses to training in endurance athletes. Metabolism. 2018 Apr;81:25-34. doi: 10.1016/j.metabol.2017.10.010. Epub 2017 Nov 3. PMID 29108901
- [Background] Zinn C, Wood M, Williden M, Chatterton S, Maunder E. Ketogenic diet benefits body composition and well-being but not performance in a pilot case study of New Zealand endurance athletes. J Int Soc Sports Nutr. 2017 Jul 12;14:22. doi: 10.1186/s12970-017-0180-0. eCollection 2017. PMID 28706467
- [Background] Burke LM, Ross ML, Garvican-Lewis LA, Welvaert M, Heikura IA, Forbes SG, Mirtschin JG, Cato LE, Strobel N, Sharma AP, Hawley JA. Low carbohydrate, high fat diet impairs exercise economy and negates the performance benefit from intensified training in elite race walkers. J Physiol. 2017 May 1;595(9):2785-2807. doi: 10.1113/JP273230. Epub 2017 Feb 14. PMID 28012184
- [Background] Paoli A, Grimaldi K, D'Agostino D, Cenci L, Moro T, Bianco A, Palma A. Ketogenic diet does not affect strength performance in elite artistic gymnasts. J Int Soc Sports Nutr. 2012 Jul 26;9(1):34. doi: 10.1186/1550-2783-9-34. PMID 22835211
- [Background] Volek JS, Freidenreich DJ, Saenz C, Kunces LJ, Creighton BC, Bartley JM, Davitt PM, Munoz CX, Anderson JM, Maresh CM, Lee EC, Schuenke MD, Aerni G, Kraemer WJ, Phinney SD. Metabolic characteristics of keto-adapted ultra-endurance runners. Metabolism. 2016 Mar;65(3):100-10. doi: 10.1016/j.metabol.2015.10.028. Epub 2015 Nov 2. PMID 26892521
- [Background] Paoli A, Rubini A, Volek JS, Grimaldi KA. Beyond weight loss: a review of the therapeutic uses of very-low-carbohydrate (ketogenic) diets. Eur J Clin Nutr. 2013 Aug;67(8):789-96. doi: 10.1038/ejcn.2013.116. Epub 2013 Jun 26. PMID 23801097